CLINICAL TRIAL: NCT02345915
Title: Evaluation of Adverse Long-term Effects in Young Adult Survivors of Acute Leukemia-LEA-JA-IPC 2014-005
Brief Title: Evaluation of Adverse Long-term Effects in Young Adult Survivors of Acute Leukemia
Acronym: LEA-JA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LEA-JA-IPC 2014-005
Record Dates: First submitted 2014-12-05; First posted 2015-01-26 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-06

CONDITIONS: Leukemia, Myeloid, Acute; Acute Lymphoid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Young adult acute leukemia-survivor (Other)
  Interventions: Other: Blood sample; Other: Electrocardiogram

INTERVENTIONS:
Other: Blood sample
Other: Electrocardiogram

SUMMARY:
Taking into account the specificities of adolescent and young adult cancer patients led agencies (in particular the French National Cancer Institute INCa, through the last Cancer Plan), to initiate projects targeting this population. Acute leukemia is among the most common cancers in adolescents and young adults. Recent therapeutic advances now allow hope for a cure in about 50% of this population. The issue of post-cancer is therefore of particular importance for young adults with cancer. Our aim is to establish the health determinants in young adult leukemia survivors and to compare the frequency of these effects and their explanatory factors to the data collected in children or adolescent leukemia survivors program (LEA). 90 patients followed up at the Institut Paoli-Calmettes cancer center and Nice University Hospital have been identified and would be included in this study.Collected data will include information on the initial disease and its treatments, physical sequelae (fertility, thyroid function, heart function, visual function, secondary tumors, viral infections, lung function, bone metabolism, iron metabolism, metabolic syndrome, osteonecrosis, alopecia ... ), quality of life, social and occupational integration and relationship with care system.

ELIGIBILITY:
Inclusion Criteria:

* Young adult (18-40 years) Leukemia survivor, in complete remission.
* Acute leukemia diagnosed since January 1980 .
* Patient Affiliated to social security or beneficiary
* Signed Informed Consent prior to any screening procedures

Exclusion Criteria:

* Emergency
* Patient unable to abide by the study protocol (for geographical, social or psychological reasons)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Late sequelae evaluation of young adult acute leukemia-survivors | 24 mois
  Main measured sequelae on: heart function, thyroid function, visual function, lung function, bone metabolism, secondary tumors, viral infections, iron metabolism, metabolic syndrome, gonadic, fertility, renal function, liver function,…
Quality-of-life assessment of young adult acute leukemia-survivors | 24 mois
  Quality of life questionnaire

SECONDARY OUTCOMES:
Comparison of the frequency of sequelae between children/adolescents (LEA cohort) and young adults acute leukemia survivors (LEA-JA) | 24 mois

CONTACTS AND LOCATIONS:
Overall Officials: Norbert VEY, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France